CLINICAL TRIAL: NCT00108667
Title: AMPA Receptor Antagonist Treatment of Parkinson's Disease
Brief Title: Talampanel to Treat Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050139; 05-N-0139
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; AMPA Antagonist; Dyskinesias; Glutamate Antagonist; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Levodopa; talampanel

INTERVENTIONS:
Drug: IV Levodopa
Drug: Talampanel

SUMMARY:
This study will evaluate the effects of the experimental drug talampanel on dyskinesias (involuntary movements) that develop in patients with Parkinson's disease as a result of long-term treatment with levodopa (Sinemet). The drug will be tested alone and in combination with amantadine-a drug commonly used to alleviate dyskinesias.

Patients between 21 and 80 years of age with Parkinson's disease and dyskinesias may be eligible for this study.

Screening and baseline evaluation. Participants are evaluated with a medical history, physical and neurologic examinations, blood and urine tests, electrocardiogram (EKG) and pregnancy test, if applicable. A chest x-ray and MRI or CT scan of the brain are done if needed. Patients stop taking all antiparkinsonian medications for one month (2 months if taking Selegiline) before the study begins and throughout its duration, except for certain medicines allowed, including Sinemet, Mirapex and Requip. Amantadine can be taken up to 1 week before beginning the study.

Dose-finding phase. Patients are admitted to the NIH Clinical Center for 2 to 3 days for a levodopa "dose-finding" procedure. For this test, patients stop taking Sinemet and instead have it infused through a vein. During the infusions, the drug dose is increased slowly until parkinsonian symptoms improve or unacceptable side effects occur or the maximum study dose is reached. Symptoms are monitored frequently. At given times during the infusion, saline is given instead of Sinemet. The infusions usually begin in the early morning and continue until evening. Patients resume taking Sinemet between infusions. (Patients who have had dosing infusions in the last 3 months do not have to undergo this phase of the study.)

After the dose-finding phase, patients are randomly assigned to take placebo (a "sugar pill") or talampanel. Those taking talampanel also receive amantadine at their usual dosages. At some point in the study, amantadine is replaced with placebo. Patients in the talampanel group also receive placebo for portions of the study.

Active study phase. At study weeks 1, 5 and 7, patients are admitted to the Clinical Center overnight for a levodopa infusion with talampanel or placebo. The day before the infusion, patients have a brief physical examination, blood and urine tests, an EKG, and a review of symptoms or changes in their condition. The next day, they receive an infusion of levodopa at the dose determined in the dose-finding phase. Then they take a pill containing either talampanel or placebo. Their parkinsonian symptoms and dyskinesias are evaluated and videotaped every 30 minutes for about 6 hours. Blood is drawn and an EKG is obtained. At the end of the infusions and ratings, patients resume their regular Parkinson's medications and are given a new supply of study medications to take home.

At weeks 2, 3, 4 and 6, patients come to the Clinical Center for a review of drug side effects. They have blood drawn and receive a new supply of study medications that last until the next visit.

Follow-up. Two weeks after the study ends, patients are contacted by phone for a review of side effects or they return to the clinic for an evaluation.

DETAILED DESCRIPTION:
Objective: to evaluate the acute effects of talampanel, a novel antagonist of AMPA type glutamate receptors, on the severity of parkinsonian signs and levodopa-associated motor response complications.

Study Population: patients with moderately advanced Parkinson's disease and dopaminergic therapy related motor complications, between the age of 21 and 80.

Study Design: randomized, controlled, proof-of-principle pilot study lasting approximately 7 weeks.

Study Outcome Parameters: the pharmacokinetic characteristics of orally administered talampanel will be measured by means of plasma drug assays, its therapeutic efficacy will be evaluated using validated motor function scales, and safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients who meet all of the following inclusion criteria on Study Day 1 will be eligible to participate in the study:

1. Between the ages of 21 and 80, inclusive;
2. Has been diagnosed with idiopathic Parkinson's disease based on the presence of a characteristic clinical history and neurologic findings;
3. Has relatively advanced disease with levodopa-associated motor response complications, including ratable peak-dose dyskinesias and wearing-off fluctuations;
4. Patient is willing to adhere to protocol requirements as evidenced by written, informed consent;
5. Patient is satisfactorily treated with levodopa with or without short acting dopamine agonist.

EXCLUSION CRITERIA:

Patients meeting any of the following exclusion criteria either at Day 0 or during the study will not be enrolled or will be immediately withdrawn from the study, as appropriate:

1. Has a history of any medical condition that can reasonably be expected to subject them to unwarranted risk, including lung disease, liver disease and clinically significant cardiac arrhythmias and/or myocardial ischemia;
2. Has clinically significant laboratory abnormalities including liver enzyme elevation; positivity to any of the autoantibodies tested at Screening (ANA, RF, anti-SM, anti-LKM)
3. Is unable to be treated with levodopa/carbidopa alone or with a single, relatively short-acting dopamine agonist, such as pramipexole or ropinirole;
4. Unable or unwilling to discontinue a prohibited concomitant medication as listed below; allowable CNS medications will be maintained at a constant dose throughout the study;
5. Has not been using an adequate contraceptive method for the last 30 days or unwilling to continue, or is not at least one year post-menopausal (if female);
6. Is pregnant or breastfeeding;
7. Is implanted with bilateral deep brain stimulators unless the stimulators are turned off during the entire study;
8. Has prior bilateral pallidotomy or other ablative surgeries for treatment of PD;
9. Has cognitive impairment (MMSE less than 25);
10. Has participated in a clinical study with an investigational drug within the last 30 days;
11. Has a condition (such as active drug or alcohol abuse) that, in the opinion of the investigators, would interfere with compliance or safety;
12. Is unwilling to sign an informed consent or to comply with protocol requirements.
13. Unilateral and bilateral pallidotomy
14. History of alcoholism.
15. Orthostatic Hypotension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-04; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kish SJ, Shannak K, Hornykiewicz O. Uneven pattern of dopamine loss in the striatum of patients with idiopathic Parkinson's disease. Pathophysiologic and clinical implications. N Engl J Med. 1988 Apr 7;318(14):876-80. doi: 10.1056/NEJM198804073181402. PMID 3352672
- [Background] Chase TN, Oh JD. Striatal mechanisms and pathogenesis of parkinsonian signs and motor complications. Ann Neurol. 2000 Apr;47(4 Suppl 1):S122-9; discussion S129-30. PMID 10762139
- [Background] Peppe A, Dambrosia JM, Chase TN. Risk factors for motor response complications in L-dopa-treated parkinsonian patients. Adv Neurol. 1993;60:698-702. No abstract available. PMID 8420213